CLINICAL TRIAL: NCT00122811
Title: The Hypertension in the Very Elderly Trial (HYVET)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Collaborators: British Heart Foundation (Other); Institut de Recherches Internationales Servier (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RG/97010
Record Dates: First submitted 2005-07-13; First posted 2005-07-22 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-08

CONDITIONS: Hypertension
Keywords: Aged; Hypertension; Stroke
MeSH Terms: conditions — Hypertension; Stroke | interventions — Perindopril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Indapamide SR 1.5mg; Perindopril 2-4mg

SUMMARY:
The purpose of this study is to assess the benefits and risks of treating very elderly (those aged 80 or older) individuals with hypertension.

DETAILED DESCRIPTION:
The benefit to risk ratio of treating hypertensives aged 80 or older has not been established. It has been suggested that at this age for each stroke prevented there is one non-stroke death. HYVET is designed to help clarify this.

HYVET is a randomised, double-blind, placebo-controlled trial in hypertensive subjects aged 80 or older. Active treatment consists of indapamide 1.5mg SR with the addition of perindopril 2mg - 4mg to reach a target blood pressure (BP) of <150/80 mmHg. Entry criteria include a systolic blood pressure of 160-199 mmHg. Patients with isolated systolic hypertension (ISH) have been recruited since August 2003.

ELIGIBILITY:
Inclusion Criteria:

* Aged 80 or older
* Sitting systolic BP 160-199 mmHg AND sitting diastolic BP < 110 mmHg

Exclusion Criteria:

* Known accelerated hypertension (retinal haemorrhages or exudates or papilloedema).
* Overt clinical congestive heart failure requiring treatment with a diuretic or angiotensin converting enzyme inhibitor. Subjects allowed if treated with digoxin only.
* Renal failure (serum creatinine of more than 150 µmol/l).
* Previous documented cerebral or subarachnoid haemorrhage in the last 6 months. (Ischaemic cerebral and cardiac events do not exclude, although the patient must be neurologically and cardiologically stable.)
* Condition expected to severely limit survival, e.g. terminal illness.
* Known secondary hypertension (e.g. renal artery stenosis, chronic renal insufficiency, and endocrine cause).
* Gout.
* Clinical diagnosis of dementia.
* Resident in a nursing home, i.e. where the dependency and care requirements of the patients are such that they require the regular input of qualified nurses and therefore the majority of staff in the home are nurses (other forms of residential care are acceptable).
* Unable to stand up or walk
* Participation in a drug trial within the past month preceding selection.
* Alcohol or drug abuse.
* Less than 2 months placebo run-in.
* Contraindications to use of trial drugs

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2000-11; Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
All strokes (fatal and non-fatal) | Duration of trial

SECONDARY OUTCOMES:
Total mortality | duration of trial
Cardiovascular mortality | Duration of trial
Cardiac mortality | Duration of trial
Stroke mortality | Duration of Trial
Fracture rates | Duration of trial

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Bulpitt, MD, FRCP, Principal Investigator — Imperial College London
Locations (7):
- Bulgaria (2):
  - Department of Internal Medicine, Clinic of Rheumatology, Plovdiv
  - University Hospital St. Anna, Sofia
- Dept of Hypertension Fu Wai Hospital, Beijing, China
- Kontinkangas Hospital Research, Oulu, Finland
- UMF Cluj, Clinica Medicala III, Cluj-Napoca, Romania
- State Scientific Research Institute of Internal Medicine, Russian Academy of Medical Sciences Siberian Department, Novosibirsk, Russia
- Imperial College London, London, United Kingdom

REFERENCES:
- [Background] Bulpitt C, Fletcher A, Beckett N, Coope J, Gil-Extremera B, Forette F, Nachev C, Potter J, Sever P, Staessen J, Swift C, Tuomilehto J. Hypertension in the Very Elderly Trial (HYVET): protocol for the main trial. Drugs Aging. 2001;18(3):151-64. doi: 10.2165/00002512-200118030-00001. PMID 11302283
- [Background] Bulpitt CJ, Peters R, Staessen JA, Thijs L, De Vernejoul MC, Fletcher AE, Beckett NS. Fracture risk and the use of a diuretic (indapamide SR) +/- perindopril: a substudy of the Hypertension in the Very Elderly Trial (HYVET). Trials. 2006 Dec 19;7:33. doi: 10.1186/1745-6215-7-33. PMID 17177983
- [Background] Peters R, Beckett N, Nunes M, Fletcher A, Forette F, Bulpitt C. A substudy protocol of the hypertension in the Very Elderly Trial assessing cognitive decline and dementia incidence (HYVET-COG) : An ongoing randomised, double-blind, placebo-controlled trial. Drugs Aging. 2006;23(1):83-92. doi: 10.2165/00002512-200623010-00008. PMID 16492072
- [Background] Pinto E, Bulpitt C, Beckett N, Peters R, Staessen JA, Rajkumar C. Rationale and methodology of monitoring ambulatory blood pressure and arterial compliance in the Hypertension in the Very Elderly Trial. Blood Press Monit. 2006 Feb;11(1):3-8. doi: 10.1097/01.mbp.0000184965.30220.10. PMID 16410734
- [Derived] Cunningham EL, Todd SA, Passmore P, Bullock R, McGuinness B. Pharmacological treatment of hypertension in people without prior cerebrovascular disease for the prevention of cognitive impairment and dementia. Cochrane Database Syst Rev. 2021 May 24;5(5):CD004034. doi: 10.1002/14651858.CD004034.pub4. PMID 34028812
- [Derived] Antikainen RL, Peters R, Beckett NS, Fagard RH, Wang JG, Rajkumar C, Bulpitt CJ. Left ventricular hypertrophy is a predictor of cardiovascular events in elderly hypertensive patients: Hypertension in the Very Elderly Trial. J Hypertens. 2016 Nov;34(11):2280-6. doi: 10.1097/HJH.0000000000001073. PMID 27552643
- [Derived] Warwick J, Falaschetti E, Rockwood K, Mitnitski A, Thijs L, Beckett N, Bulpitt C, Peters R. No evidence that frailty modifies the positive impact of antihypertensive treatment in very elderly people: an investigation of the impact of frailty upon treatment effect in the HYpertension in the Very Elderly Trial (HYVET) study, a double-blind, placebo-controlled study of antihypertensives in people with hypertension aged 80 and over. BMC Med. 2015 Apr 9;13:78. doi: 10.1186/s12916-015-0328-1. PMID 25880068
- [Derived] Peters R, Beckett N, Pereira L, Poulter R, Pinto E, Ma S, Dumitrascu D, Barrowdale D, Butler M, Fletcher A, Bulpitt C. The clock drawing test, mortality, incident cardiovascular events and dementia. Int J Geriatr Psychiatry. 2015 Apr;30(4):416-21. doi: 10.1002/gps.4153. Epub 2014 Jun 12. PMID 24920166
- [Derived] Antikainen RL, Beckett N, Peters R, Fagard R, Rajkumar C, Wang J, Stoyanovsky V, Barrowdale D, Bulpitt CJ; HYVET Study Group. Prevalence and covariates of electrocardiographic left ventricular hypertrophy in the Hypertension in the Very Elderly Trial. J Hypertens. 2013 Jun;31(6):1224-32. doi: 10.1097/HJH.0b013e32836040a4. PMID 23588194
- [Derived] Peters R, Beckett N, Poulter R, Burch L, Narkiewicz K, Fagard R, Nitsch D, Wang N, Li M, Fletcher A, Bulpitt C. Kidney function in the very elderly with hypertension: data from the hypertension in the very elderly (HYVET) trial. Age Ageing. 2013 Mar;42(2):253-8. doi: 10.1093/ageing/afs109. Epub 2012 Aug 21. PMID 22910302
- [Derived] Beckett N, Peters R, Tuomilehto J, Swift C, Sever P, Potter J, McCormack T, Forette F, Gil-Extremera B, Dumitrascu D, Staessen JA, Thijs L, Fletcher A, Bulpitt C; HYVET Study Group. Immediate and late benefits of treating very elderly people with hypertension: results from active treatment extension to Hypertension in the Very Elderly randomised controlled trial. BMJ. 2011 Jan 4;344:d7541. doi: 10.1136/bmj.d7541. PMID 22218098
- [Derived] Peters R, Beckett N, Burch L, de Vernejoul MC, Liu L, Duggan J, Swift C, Gil-Extremera B, Fletcher A, Bulpitt C. The effect of treatment based on a diuretic (indapamide) +/- ACE inhibitor (perindopril) on fractures in the Hypertension in the Very Elderly Trial (HYVET). Age Ageing. 2010 Sep;39(5):609-16. doi: 10.1093/ageing/afq071. Epub 2010 Jun 23. PMID 20573778
- [Derived] Peters R, Pinto E, Beckett N, Swift C, Potter J, McCormack T, Nunes M, Grimley-Evans J, Fletcher A, Bulpitt C. Association of depression with subsequent mortality, cardiovascular morbidity and incident dementia in people aged 80 and over and suffering from hypertension. Data from the Hypertension in the Very Elderly Trial (HYVET). Age Ageing. 2010 Jul;39(4):439-45. doi: 10.1093/ageing/afq042. Epub 2010 May 23. PMID 20497949
- [Derived] Peters R, Beckett N, Forette F, Tuomilehto J, Ritchie C, Walton I, Waldman A, Clarke R, Poulter R, Fletcher A, Bulpitt C. Vascular risk factors and cognitive function among 3763 participants in the Hypertension in the Very Elderly Trial (HYVET): a cross-sectional analysis. Int Psychogeriatr. 2009 Apr;21(2):359-68. doi: 10.1017/S1041610208008302. Epub 2009 Feb 27. PMID 19250558
- [Derived] Peters R, Beckett N, Forette F, Tuomilehto J, Clarke R, Ritchie C, Waldman A, Walton I, Poulter R, Ma S, Comsa M, Burch L, Fletcher A, Bulpitt C; HYVET investigators. Incident dementia and blood pressure lowering in the Hypertension in the Very Elderly Trial cognitive function assessment (HYVET-COG): a double-blind, placebo controlled trial. Lancet Neurol. 2008 Aug;7(8):683-9. doi: 10.1016/S1474-4422(08)70143-1. Epub 2008 Jul 7. PMID 18614402
- [Derived] Beckett NS, Peters R, Fletcher AE, Staessen JA, Liu L, Dumitrascu D, Stoyanovsky V, Antikainen RL, Nikitin Y, Anderson C, Belhani A, Forette F, Rajkumar C, Thijs L, Banya W, Bulpitt CJ; HYVET Study Group. Treatment of hypertension in patients 80 years of age or older. N Engl J Med. 2008 May 1;358(18):1887-98. doi: 10.1056/NEJMoa0801369. Epub 2008 Mar 31. PMID 18378519